CLINICAL TRIAL: NCT00440700
Title: Reducing Sedative Exposure in Ventilated ICU Patients
Brief Title: Anxiety Self-Management for ICU Patients Receiving Mechanical Ventilation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0601M79066
Record Dates: First submitted 2007-02-23; First posted 2007-02-27 (Estimated); Results first posted 2013-04-26 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Anxiety
Keywords: Ventilator; chronic obstructive pulmonary disease; Anxiety
MeSH Terms: conditions — Anxiety Disorders; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Patient-directed music (Experimental): Patients select preferred music for listening through headphones whenever they like for as long as they like whenever feeling anxious, desire some rest and quiet time, or for listening enjoyment while mechanically ventilated in the ICU.
  Interventions: Behavioral: Anxiety Self-Management, Patient preferred relaxing music
- Headphones (Active Comparator): Noise-canceling headphones only (no music) are applied by the patient to block out noise/sound in the ICU whenever desired.
  Interventions: Behavioral: Control 1: Noise-cancelling headphones
- Standard of Care (Other): Patients receive usual care for the ICU and are encouraged to self-initiate rest periods twice daily.
  Interventions: Behavioral: Control 2: Standard of Care

INTERVENTIONS:
Behavioral: Anxiety Self-Management, Patient preferred relaxing music — Experimental group randomized to patient-directed music intervention where subjects listened to tailored, self-selected music as desired (frequency and length determined by the individual subject) each day they are receiving mechanical ventilatory support.
  Other Names: self-initiated music listening
  Arms: Patient-directed music
Behavioral: Control 1: Noise-cancelling headphones — Control group: noise-canceling headphones only where subjects wear headphones as desired (frequency and length determined by the individual subject) each day they are receiving mechanical ventilatory support.
  Other Names: noise-reduction headphones
  Arms: Headphones
Behavioral: Control 2: Standard of Care — Usual ICU nursing care.
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to test whether patients who are receiving mechanical ventilation in the ICU who listened to preferred, relaxing music whenever they desire for as long as they desire will have less anxiety, receive fewer medications, stay in the ICU for a shorter time, and experience less stress than patients who do not listen to music.

DETAILED DESCRIPTION:
A three group randomized trial with repeated measures. Participants are assigned by chance to one of three groups: 1) patient-directed, as desired music listening through headphones, 2) noise-canceling headphones only, or 3) usual care. Participants remain in the study, up to 30 days, as long as they are receiving mechanical ventilation in the ICU, choose to withdraw, or become unable to complete the daily anxiety assessments. Information is collected daily on patient-perceived anxiety levels (visual analog scale & State Anxiety Inventory), ventilator settings, and all medications received. Urine is collected each day the participant is on the ventilator to determine level of stress (cortisol) if the kidneys are functioning appropriately and the participant is not receiving medications known to influence cortisol levels.

Mechanical ventilation is a common treatment for respiratory problems for patients in the ICU. Patients receiving mechanical ventilation experience much anxiety and distress from the placement of the endotracheal tube (breathing tube) and the mechanical ventilator itself. The usual treatment for these symptoms are medications, which are very potent and have numerous adverse side effects, removing patient involvement and control from managing these symptoms. Music has been shown to decrease anxiety and promote relaxation in limited, single listening intervention studies with patients in the ICU on ventilators. This study tests whether having patients listen to preferred music (familiar & comforting) whenever feeling anxious and wanting to relax for as long as they would like to listen to music through headphones throughout the entire time they are on the ventilator can improve outcomes such as less anxiety, shorter time on the ventilator, receipt of fewer medications, and less stress when compared to patients who do not listen to music while they are on the ventilator. Results from this study will advance nursing science by providing evidence on the efficacy of a simple, self-directed intervention that the millions of patients who receive mechanical ventilation each year in the ICU can use themselves to treat the very common symptoms of anxiety and distress. Results from this study will expand the knowledge base of adjunctive interventions that can be implemented in the ICU to involve patients directly in managing their own symptoms, ultimately improving patient outcomes.

Patients who are alert and can provide consent are invited to participate if they are on the ventilator in one of the participating ICUs. Patients remain in the study for as long as they are on the ventilator (up to 30 days) and can provide daily assessment of their anxiety levels. Patients are free to withdraw, however, at any time. Patients randomized to music receive an assessment of their music preferences by a professional music therapist. The music therapist then develops a music collection for each participant, based in individual preferences, that is kept at the bedside throughout the duration of being on the ventilator. The music therapist also visits with music participants' daily to determine if preferences have changed and if he/she desires additional music compact disks (CDs) to be kept at the bedside. Data is collected from the medical record on all medications and ventilator settings each day the participant is enrolled in the study. All urine is collected each day the participant remains in the study if the kidneys are functioning properly and the participant is not receiving medications known to influence cortisol, a marker for an integrative level of stress.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who is alert, on the ventilator because there is some condition involving the lungs preventing him/her from breathing on his/her own and willing and able to provide own consent.

Exclusion Criteria:

* On the ventilator because of a surgical procedure, not alert and unable to provide own consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2006-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Chlan, PhD, RN, Principal Investigator — University of Minnesota School of Nursing
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Heiderscheit A, Johnson K, Chlan LL. Analysis of Preferred Music of Mechanically Ventilated Intensive Care Unit Patients Enrolled in a Randomized Controlled Trial. J Integr Complement Med. 2022 Jun;28(6):517-529. doi: 10.1089/jicm.2021.0446. Epub 2022 Apr 4. PMID 35377238
- [Derived] Chlan LL, Heiderscheit A, Skaar DJ, Neidecker MV. Economic Evaluation of a Patient-Directed Music Intervention for ICU Patients Receiving Mechanical Ventilatory Support. Crit Care Med. 2018 Sep;46(9):1430-1435. doi: 10.1097/CCM.0000000000003199. PMID 29727366
- [Derived] Chlan LL, Weinert CR, Heiderscheit A, Tracy MF, Skaar DJ, Guttormson JL, Savik K. Effects of patient-directed music intervention on anxiety and sedative exposure in critically ill patients receiving mechanical ventilatory support: a randomized clinical trial. JAMA. 2013 Jun 12;309(22):2335-44. doi: 10.1001/jama.2013.5670. PMID 23689789

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care: Patients receive usual care for the ICU and are encouraged to self-initiate rest periods twice daily.
Period: Overall Study
Arm/Group | Patient-directed Music | Headphones | Usual Care
Started | 122 | 118 | 124
Completed | 114 | 110 | 120
Not Completed | 8 | 8 | 4
Not completed — Withdrawal by Subject | 8 | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient-directed Music | Headphones | Usual Care | Total
Number analyzed (Participants) | 122 | 118 | 124 | 364
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 88 | 90 | 95 | 273
  >=65 years | 34 | 28 | 29 | 91
Age Continuous [Mean (Standard Deviation); unit: years] | 60.4 (15.4) | 59.4 (14.3) | 57.8 (13.5) | 59.2 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 54 | 68 | 188
  Male | 56 | 64 | 56 | 176
Region of Enrollment [Number; unit: participants]
  United States | 122 | 118 | 124 | 364

OUTCOME MEASURES:

1. Primary Outcome: Sedative Exposure
Description: Sedative exposure was measured by: 1) the number (dose frequency) of sedative medication doses administered in a 4-hour time period each day and 2) by an aggregate dose intensity of sedative medications administered in a 4-hour time period each day based on all subjects receiving sedative medications on any individual study day yielding a sedation intensity score. A sedation intensity score was calculated for each study group each study protocol day, up to 30 days. Higher sedation intensity scores indicate more sedative exposure. If a subject did not receive any sedation, the sedative exposure score is zero for that respective day.
Time Frame: Daily up to 30 days
Population: Participants with 2 or more days of study enrollment data were included in the analysis for this aim.
Measure: Median (Full Range); unit: exposures/4-hours per day
Arm/Group | Patient-directed Music | Headphones | Usual Care
Number analyzed (Participants) | 87 | 90 | 89
exposures/4-hours per day | 1 [0 to 12] | 7 [0 to 10] | 6 [0 to 12]

2. Primary Outcome: State Anxiety
Description: Participants reported their current level of anxiety each day enrolled in the study in response to the question "how are you feeling today"/ The Visual analog scale-anxiety was used to evaluate the self-report of anxiety. Scores range from 0 = not anxious at all to 100 = the most anxious ever. Higher numbers indicate greater anxiety. Daily anxiety scores from all subjects were combined and analyzed for each group resulting in an overall mean anxiety score at the end of the study protocol of 30 days.
Time Frame: Daily up to 30 days
Population: Participants with 3 or more visual analog scale-anxiety ratings were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient-directed Music | Headphones | Usual Care
Number analyzed (Participants) | 86 | 81 | 74
units on a scale | 40 (32.4) | 59 (30.1) | 55 (29.7)
Statistical Analysis 1: Comparison: Patient-directed Music vs Headphones vs Usual Care; Mixed models analysis was used to determine if there were any differences in anxiety levels in patients who listen to music as compared to headphones only or usual ICU care; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Slope = 15.5

3. Secondary Outcome: Length of ICU Stay
Description: Length of ICU stay was measured in days from the first day participant was admitted to the unit until discharged, transferred, or died in the ICU. This was the total time that any participant was in the intensive care unit which could have been longer than the 30 study protocol .
Time Frame: From date of ICU admission to extubation or discharge or date of death from any cause, whichever came first assessed up to 60 days
Population: The number of participants includes all of those patients who were enrolled into the study protocol, regardless of their length of study participation.
Measure: Mean (Standard Error); unit: days
Arm/Group | Patient-directed Music | Headphones | Usual Care
Number analyzed (Participants) | 122 | 118 | 124
days | 18.8 (.85) | 19.3 (.87) | 18.7 (.85)

4. Secondary Outcome: Length of Mechanical Ventilatory Support
Description: Length of mechanical ventilatory support was defined as the number of days from initial intubation and placement on mechanical ventilation to the day of extubation or death for participants in each group.
Time Frame: From initial intubation date to extubation or death, whichever came first, assessed up to 30 days.
Population: Includes all subjects enrolled regardless of length of protocol participation. Mean number of days mechanically ventilated was calculated for the subjects randomized to each group/arm.
Measure: Mean (Standard Error); unit: days
Arm/Group | Patient-directed Music | Headphones | Usual Care
Number analyzed (Participants) | 122 | 118 | 124
days | 4.4 (.61) | 5.8 (.62) | 5.9 (.60)
Statistical Analysis 1: Comparison: Patient-directed Music vs Usual Care; Length of mechanical ventilatory support was assessed among all 3 groups. Usual usual care was the reference group as compared to the experimental patient-directed music group; Test type: Superiority or Other; p < 0.05, Kruskal-Wallis; Mean Difference (Final Values) = 1.5, Standard Error of Mean 0.61 — Usual care was the reference comparison group

5. Secondary Outcome: Urinary Cortisol
Description: Stress was measured by the biomarker urinary cortisol. 24-hour urine collections were obtained from eligible participants who were not receiving steroids or other medications known to affect cortisol and who had intact renal function. 24-hour urinary cortisol results were used as an integrative measure of stress (mg/day).
Time Frame: Daily up to 30 days
Population: All participants with functioning kidneys who were not receiving steroids or other medications known to affect cortisol and who had two or more 24-hour urine collections were included in the analysis.
Measure: Median (Full Range); unit: total milligrams per day
Arm/Group | Patient-directed Music | Headphones | Usual Care
Number analyzed (Participants) | 19 | 27 | 19
total milligrams per day | 29.3 [1 to 181.4] | 54 [8.8 to 241] | 33 [5.9 to 264.8]
Statistical Analysis 1: Comparison: Patient-directed Music vs Headphones vs Usual Care; Cortisol levels were compared among all 3 groups; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Slope = 5

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Patient-directed Music | Headphones | Usual Care
Serious Adverse Events (participants affected / at risk) | 5/122 | 5/118 | 7/124
Other Adverse Events (participants affected / at risk) | 0/122 | 1/118 | 1/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patient-directed Music (N=122) | Headphones (N=118) | Usual Care (N=124)
Self-extubation (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5) | 5 (5)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure activity (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) — seizure activity noted in patient after ICU admission for stroke
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patient-directed Music (N=122) | Headphones (N=118) | Usual Care (N=124)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) — Subject noted to have history of allergies. Ears became stuffy after wearing study headphones.
Impaired hearing (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) — New loss of hearing acuity; determined to be of unknown etiology after ear, nose throat consult. No issues with understanding verbal communication with staff or research staff.

LIMITATIONS AND CAVEATS:
Overall limitations of the trial include the challenges of obtaining informed consent from patients' themselves. Many times patients were too sedated or not alert enough to participate in the consent process.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No